CLINICAL TRIAL: NCT07163273
Title: Monthly Alternating NALIRIFOX and GnP in the First-Line Setting for Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0950
Record Dates: First submitted 2025-07-14; First posted 2025-09-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Fluorouracil; Leucovorin; Oxaliplatin; irinotecan sucrosofate; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NALIRIFOX (Active Comparator): NALIRIFOX consists of 5-FU 2400 mg/m2 over 46 hours, liposomal irinotecan 50 mg/m2, and oxaliplatin 60 mg/m2, which would be given on Day 1 and Day 15
  Interventions: Drug: NALIRIFOX
- Gemcitabine plus nab-Paclitaxel (GnP) (Active Comparator): GnP consists of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2, given on Days 1, 8, and 15.
  Interventions: Drug: Gemcitabine plus nab-Paclitaxel (GnP)

INTERVENTIONS:
Drug: NALIRIFOX — NALIRIFOX consists of 5-FU 2400 mg/m2 over 46 hours, liposomal irinotecan 50 mg/m2, and oxaliplatin 60 mg/m2, which would be given on Day 1 and Day 15
  Other Names: 5fu/ leucovorin / oxaliplatin / liposomal irinotecan
  Arms: NALIRIFOX
Drug: Gemcitabine plus nab-Paclitaxel (GnP) — GnP consists of gemcitabine 1000 mg/m2 and nab-paclitaxel 125 mg/m2, given on Days 1, 8, and 15.
  Other Names: Gemcitabine/nab-Paclitaxel
  Arms: Gemcitabine plus nab-Paclitaxel (GnP)

SUMMARY:
A prospective, interventional, single-center, single-arm, open-label, phase II study for patients with metastatic pancreatic cancer. The intervention consists of monthly alternating standard chemotherapy regimens-NALIRIFOX and GnP. The hypothesis is that induction therapy with alternating NALIRIFOX and GnP has better efficacy compared to historical observation.

ELIGIBILITY:
Inclusion:

* >18 years of age
* Histologically proven pancreatic ductal adenocarcinoma, poorly differentiated carcinoma, or adenosquamous carcinoma
* Radiographic evidence of metastatic disease
* At least 1 measurable target lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Metastatic relapse of previously resected pancreatic cancer is allowed provided the patient is more than 6 months from last SOC adjuvant treatment
* ECOG PS 0-1
* Laboratory assessments within 14 days as indicated below:

  * Hemoglobin > 9.0 g/dL (patients with hemoglobin < 9 g/dL may be transfused prior to study enrollment)
  * Platelet count > 100 x 10^9/L
  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  * Total bilirubin < 3 x upper limit of normal (ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x ULN (if liver metastases are present, AST and ALT < 5 x ULN is permitted.
  * Creatinine ≤1.5 ULN
  * Creatinine clearance > 40 mL/min as calculated by Cockcroft-Gault formula
  * APTT (aPTT) ≤ 1.5 × ULN. For subjects receiving unfractionated heparin < 2.5 × ULN, or within acceptable range considered by the investigator.
  * PT/INR INR ≤ 1.5 × ULN. For subjects receiving warfarin, 2.0 -3.0, or within acceptable range considered by the investigator.
* Women of childbearing potential must be surgically sterile or postmenopausal or must have a negative pregnancy test (serum or urine) prior to study enrolment and must use effective barrier contraception or abstinence during the treatment period. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions and therefore are not considered effective for this study. Male patients must be surgically sterile or use effective contraception or abstinence during the treatment period. The definition of effective contraception will be based on investigator discretion. Female and male patients are advised to use effective contraceptives for at least 9 months after the last treatment dose.
* Ability to understand and willing to sign informed consent form

Exclusion:

* A history of other disease, metabolic dysfunction, physical examination finding or clinical laboratory test result suspicious of a disease or condition which, in the opinion of the investigator, would compromise patient safety due to risk of treatment complications or could affect interpretation of the study results
* Ampullary, acinar, squamous, and neuroendocrine histology
* Presence of central nervous system metastases
* Life expectancy < 12 weeks
* Pregnant or breastfeeding women
* Prior neuropathy > grade 1 as per CTCAE v5
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Major surgery within 4 weeks prior to initiation of the study treatment, without full recovery
* Any past chemotherapy delivered for metastatic pancreatic cancer
* Known somatic or germline mutations in BRCA1, BRCA2, or PALB2
* Active second malignancy whose prognosis has a high likelihood of impacting survival
* Any other medical or social condition deemed by the investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results. Patients also unwilling or unable to comply with study procedures and/or study visits, including long-term follow-up for survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Determine 6-month Progression Free Survival (PFS) | 6 months
  The primary endpoint is 6-month PFS rate defined as the proportion of patients alive and progression free (by RECIST v.1.1) at 6 months after treatment initiation. PFS events will be classified as either local progression, distant recurrence, secondary malignancy, or death.

SECONDARY OUTCOMES:
Overall Response Rate | 24 months
  Overall response rate, defined as the proportion of patients whose best response is partial response or complete response by RECIST v.1.1
Disease Control Rate | 24 months
  Disease control rate, defined as the proportion of patients whose best response is stable disease, partial response, or complete response, by RECIST v.1.1
Overall Survival | 24 months
  OS, defined as the time from treatment initiation to death. Patients living without disease progression will be censored at the date of last assessment
Determine Toxicities using the NCI CTCAE v. 5.0 | 24 months
  AEs will be monitored, and the incidence, severity, and relationship to study drug will be reported.
Time to Treatment Failure | 24 months
  Time to treatment failure, defined as the time from treatment initiation to discontinuation of treatment, either due to progression or intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg Cancer Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No